CLINICAL TRIAL: NCT07083895
Title: Empowering Cardiovascular Health in Custodial Grandparents
Acronym: ECG
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, MinKyoung Song, Associate Professor, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: STUDY00028858
Record Dates: First submitted 2025-07-02; First posted 2025-07-24 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Cardiovascular Disease (CVD) Risk Factors
Keywords: Rural Caregiver Heart Health Education (RICHH); Custodial grandparents; Grandparent caregivers; Cardiovascular disease (CVD) risk factors; Community health workers; Grandchildren
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Modified RICHH Intervention (Experimental): The investigators will employ a re-designed RICHH intervention and determine its feasibility and acceptability with custodial grandparents.
  Interventions: Behavioral: Modified RICHH
- Standard of Care (Active Comparator): The usual care control group will receive mini-iPads loaded with Caregiver and CVD risk reduction pamphlets in PDF format along with the associated links from the American Heart Association. Because the investigators may identify CVD risk factors in baseline testing in participants who do not know they have them, it would be unethical not to provide at least usual standard of care for these. Thus, all individuals enrolled in the study and in whom the investigators identify CVD risk factors will receive referral to a primary care provider for management of the CVD risk factors identified.
  Interventions: Behavioral: Standard of Care (SOC)

INTERVENTIONS:
Behavioral: Modified RICHH — The RICHH intervention is an educational-behavioral and counseling intervention that promotes caregivers' knowledge, skills and motivation to engage in CVD risk reduction. The intervention is delivered individually to caregivers in their homes using video-conferencing technology on mini-iPads. The program consists of 12 weekly sessions [30-45 minutes] that will be held at the caregivers' preferred times. RICHH consists of 6 interactive modules (i.e., self-management for heart health, depressive symptom management, heart healthy eating, physical activity, co-morbid condition management, and adherence to medication and smoking cessation).
  The modified RICHH intervention utilizes focus group outcomes to employ modifications needed to target custodial grandparents from varied backgrounds (e.g., high ACEs, SDoH groups).
  Arms: Modified RICHH Intervention
Behavioral: Standard of Care (SOC) — Referral to primary care provider
  Other Names: Usual Care
  Arms: Standard of Care

SUMMARY:
In this study, the investigators will tailor an existing intervention (Rural Caregiver Heart Health Education (RICHH)) protocol and test its feasibility, acceptability, and initial effect with grandparent caregivers.

ELIGIBILITY:
Grandparent (inclusion):

* Provides full-time care to at least one grandchild (< 18 years old) for at least 6 months, with no biological parent residing in the household or providing substantial care to the children
* Lives in Oregon
* Has English proficiency sufficient for informed consent and completion of study measures
* Provides signed informed consent

Grandparent (exclusion)

* Plans for transfer of care to other caregivers or setting for the next 12 months
* Has significant physical or emotional impairment, or psychiatric illness that might interfere with engagement in their own self-management or that is likely to result in their needing a caregiver in the next 12 months
* Chronic drug abuse
* Current active cancer (i.e., undergoing active treatment for cancer) other than isolated skin cancer

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2028-01-31 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants who complete the intervention and follow-up | 4 months after baseline and 6 months after baseline
  Feasibility is measured by the count of participants who complete the intervention and follow-up components of the study
Percentage of participants who indicate acceptability of study intervention | 4 months after baseline
  Acceptability will be assessed in the domains of affective attitude, burden, opportunity costs, perceived effectiveness, and self-efficacy
Physical activity | At baseline, 4 months after baseline, and 6 months after baseline
  Measured using ActiGraph GT9X Link devices. The ActiGraph algorithms generate accurate and reliable data on total energy expenditure (kcal/day). Participants will wear the devices over 7-day periods at each data collection point. For each participant, the average proportion of time per day in moderate-to-vigorous physical activity (MVPA), out of total time wearing the monitors, will be calculated.
Food intake | At baseline, 4 months after baseline, and 6 months after baseline
  Measured using the self-report Viocare Food Frequency Questionnaire. Data from Viocare will be used to generate Healthy Eating Index scores, which range from 0 to 100. Higher scores indicate better dietary quality.
Body mass index | At baseline, 4 months after baseline, and 6 months after baseline
  BMI (kg/m2) will be calculated from height and body weight measured

SECONDARY OUTCOMES:
Blood pressure | At baseline, 4 months after baseline, and 6 months after baseline
  Measured by the average of three consecutive resting blood pressure measurements (both systolic and diastolic pressures).
Lipids | At baseline, 4 months after baseline, and 6 months after baseline
  Measured using non-fasting total cholesterol obtained via finger stick
Hemoglobin A1c (HbA1c) | At baseline, 4 months after baseline, and 6 months after baseline
  Measured using non-fasting HbA1c obtained via finger stick
Nicotine exposure | At baseline, 4 months after baseline, and 6 months after baseline
  Assessed via self-report of cigarette use/inhaled nicotine use, or secondhand smoke exposure. AHA Life's Essential 8 algorithm will generate a score (0-100), with lower scores indicating greater risk.
Depressive symptoms | At baseline, 4 months after baseline, and 6 months after baseline
  Depressive symptoms will be assessed using the Patient Health Questionnaire-9 (PHQ-9). Scores range from 0 to 27, with higher scores indicating more severe depressive symptoms.
Waist circumference | At baseline, 4 months after baseline, and 6 months after baseline
  Waist circumference will be measured using a nonextensible tape. At least two independent measurements will be taken and averaged.

CONTACTS AND LOCATIONS:
Overall Officials: MinKyoung Song, PhD, RN, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: Yes